CLINICAL TRIAL: NCT05809089
Title: Early-initiated High Flow Nasal Oxygen Therapy in Pneumonia Patients Presenting With Acute Hypoxemic Respiratory Failure
Brief Title: HFNO in Pneumonia Patients Presenting With Acute Hypoxemic Respiratory Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Doaa Magdy Eid, associate proffessour, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 04355751
Record Dates: First submitted 2023-03-06; First posted 2023-04-12 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Pneumonia
MeSH Terms: conditions — Pneumonia | interventions — Noninvasive Ventilation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- (High flow nasal cannula (HFNC) (Active Comparator): This arm should have the intervention"High flow nasal cannula (HFNC)" assigned to it.
  Interventions: Device: High flow nasal cannula (HFNC)
- Noninvasive ventilation (NIV) (Active Comparator): This arm should have the intervention "Noninvasive ventilation (NIV)" assigned to it.
  Interventions: Device: Noninvasive ventilation (NIV)

INTERVENTIONS:
Device: High flow nasal cannula (HFNC) — High-flow nasal cannula device was utilized. Humidifier temperature was set at 37°C via large-bore bi-nasal prongs, and inspired oxygen (FiO2) was adjusted to maintain oxygen saturation by pulse oximetry (SpO2) ≥ 90%.The flow was initially set at 10 L/min and titrated upward in 5 L/min steps until patients experienced discomfort.
  Patient will be evaluated every 8 hours and discontinued the device for eating, drinking and coughing up secretion and returned back to the device for 72 hours.
  Arms: (High flow nasal cannula (HFNC)
Device: Noninvasive ventilation (NIV) — Patients initiated NIV; Inspiratory positive airway pressure (IPAP) was initiated at 10-12 cmH2O, and expiratory positive airway pressure (EPAP) started at 4-5 cmH2O. FIO2 was adjusted to maintain SpO2 ≥ 90%. The same protocol as done in HFNC, patient will be evaluated every 8 hours and discontinued the device and returned back to the device for re- evaluation within 72 hours
  Arms: Noninvasive ventilation (NIV)

SUMMARY:
High-flow nasal oxygen (HFNO) therapy is an upcoming and beneficial modality for patients with acute hypoxemic respiratory failure (AHRF).

To evaluate whether early use of HFNO in pneumonia patients with (AHRF) can reduce the need for invasive ventilation.

DETAILED DESCRIPTION:
* Pneumonia adults patients (age>18 years) with AHRF were eligible for this study after conventional oxygen therapy failure.
* The criteria for diagnosing AHRF were defined as the presence of a respiratory rate (RR) more than 25 breaths/min with SpO2 less than 92%, and/or the arterial oxygen partial pressure (PaO2) to FiO2 ratio less than 300 mmHg while breathing oxygen delivered by a conventional venturi device at a fraction of inspiration oxygen of 0.5 (as per maximum for Venturi mask) administered for at least 60 minutes.

Eligible patients were randomized to receive either HFNO or NIV respiratory support throughout the hospitalization period. Randomization was stratified by a laboratory scientist not involved in the study using the technique of shuffled sealed envelopes.

ELIGIBILITY:
Inclusion Criteria:

* Pneumonia adults patients (age>18 years) with AHRF were eligible for this study after conventional oxygen therapy failure.
* The criteria for diagnosing AHRF were defined as the presence of a respiratory rate (RR) more than 25 breaths/min with SpO2 less than 92%, and/or the arterial oxygen partial pressure (PaO2) to FiO2 ratio less than 300 mmHg while breathing oxygen delivered by a conventional venturi device at a fraction of inspiration oxygen of 0.5 (as per maximum for Venturi mask) administered for at least 60 minutes.

Exclusion criteria:

* Patients requiring emergency intubation,
* Recent esophageal, facial, or cranial trauma or surgery,
* Severely decreased consciousness (Glasgow coma scale [GCS] of 11 or less),
* Severe hemodynamic instability (patient on inotropic or vasopressor support), ° Severe ventricular arrhythmia or myocardial ischemia,
* Tracheotomy or other upper airway disorders,
* Active upper gastrointestinal bleeding, and
* Inability to clear respiratory secretions .

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2020-11-20 (Actual); Primary Completion 2023-01-20 (Actual); Study Completion 2023-02-20 (Actual)

PRIMARY OUTCOMES:
The rate of intubation among participant | within 72 hours after admission
  The criteria for immediate intubation were: cardiac arrest or obvious hemodynamic instability, refractory hypoxemia (PaO2 < 50mmHg with sufficient oxygen therapy), significant hypercapnia with pH ≤ 7.20, loss of consciousness or gasping for air, psychomotor agitation, or severe dyspnea (respiratory frequency > 40/min)

SECONDARY OUTCOMES:
Improvement of respiratory exchanges compared to baseline | hospital admission until the achievement of clinical stability (72 hours)
  Evaluation of oxygenation (paO2 in mmHg )and hypercapnea (Pa Co2 in mmHg )using arterial blood gas )
Dyspnea | hospital admission until the achievement of clinical stability (72 hours)
  Borg dyspnea scale
Mortality rate | at 28 days
  Patient died after reintubation

CONTACTS AND LOCATIONS:
Overall Officials: ahmed metwaly, dectorate, Principal Investigator — Assiut University
Locations (1):
- Doaa Magdy Eid, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Magdy DM. Outcome of Early Initiation of High-flow Nasal Oxygen Therapy among Pneumonia Patients Presenting with Acute Hypoxemic Respiratory Failure. Indian J Crit Care Med. 2024 Aug;28(8):753-759. doi: 10.5005/jp-journals-10071-24769. Epub 2024 Jul 31. PMID 39239186